CLINICAL TRIAL: NCT05506176
Title: A Multicenter, Randomized, Double-blind, Phase Ⅱ/Ⅲ Clinical Study to Evaluate the Efficacy and Safety of SIM0417 Orally Co-Administered With Ritonavir in Symptomatic Adult Participants With Mild to Moderate COVID-19
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of SIM0417 Orally Co-Administered With Ritonavir in Symptomatic Adult Participants With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0417-301
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Mild to Moderate COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SIM0417

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIM-0417 (Experimental): orally administrated SIM0417+ ritonavir
  Interventions: Drug: SIM0417
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SIM0417 — dose of 750 mg SIM0417 with 100 mg ritonavir.
  Other Names: Simnotrelvir
  Arms: SIM-0417
Drug: Placebo — Placebo (tablet)
  Arms: Placebo

SUMMARY:
This Phase Ⅱ/Ⅲ study is to evaluate whether or not there is a difference in time recovery of COVID-19 signs and symptoms through Day 29 between SIM0417/ritonavir and placebo.

DETAILED DESCRIPTION:
The efficacy, safety, and tolerability of SIM0417/ritonavir compared to placebo will be investigated. The exposure to SIM0417 in this population will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years of age (or the minimum country-specific age of consent if >18) at the time of signing the informed consent/assent form.
2. Initial positive SARS-CoV-2 tested by RT-PCR or rapid antigen test within 5 days (120 h) prior to the first dose of study drug collected from any respiratory tract specimen (e.g., oropharyngeal, NP or nasal swab, or saliva).
3. Initial onset of signs/symptoms attributable to COVID-19 within 3 days prior to the day of the first dose of study drug. The onset time of symptoms was defined as the time when body temperature first rose; or the onset of any of these COVID-19 symptoms.
4. At least one of the following symptoms of COVID-19 present within 24 hours prior to the first dose of study drug and meeting severity.
5. Has mild or moderate COVID-19.
6. Participants agree to take highly effective contraceptive measures from signing the informed consent to at least 1 month after the last dose of study intervention.
7. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
8. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent.

Exclusion Criteria:

1. Urgent or expected need for nasal high-flow oxygen therapy or positive pressure ventilation, invasive mechanical ventilation or Extracorporeal membrane oxygenation(ECMO).
2. Known medical history of active liver disease (other than nonalcoholic hepatic steatosis), including acute or chronic active hepatitis B or C infection, primary biliary cirrhosis, Child-Pugh Class B or C, or acute liver failure.
3. Receiving dialysis or have known moderate to severe renal impairment (ie, eGFR <45 mL/min/1.73 m2 within 6 months of the screening visit, using the serum creatinine-based CKD-EPI formula).
4. Compromised immune system (including patients receiving long-term immunosuppressant therapy, or those with progressed or relapsed cancer or human immunodeficiency virus [HIV] infection).
5. Moderate to severe congestive heart failure (New York Heart Association class III or IV) within 6 months prior to Screening, recent (within the past 6 months prior to Screening) cerebrovascular accident, myocardial infarction, coronary artery stenting, or uncontrolled hypertension (defined as documented systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg).
6. Acute episode of chronic respiratory diseases, including bronchial asthma, chronic obstructive pulmonary disease.
7. Suspected or confirmed concurrent active systemic infection other than COVID-19 (eg, co-infected with influenza) that may interfere with the evaluation of response to the study intervention.
8. Any comorbidity requiring surgery within 14 days prior to study entry, or that is considered life-threatening within 30 days prior to study entry, as determined by the investigator.
9. Has hypersensitivity or other contraindication to any of the components of the study interventions.
10. Other medical or psychiatric conditions including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
11. Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥30 per minute, heart rate ≥125 per minute, oxygen saturation (SpO2) of ≤93% on room air or the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) <300 obtained at rest within 24 hours prior to randomization.
12. Treatment with antivirals against SARS-CoV-2 within 14 days prior to the first dose of randomization.
13. Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance and for which elevated plasma concentrations may be associated with serious and/or life-threatening events during study treatment and for 4 days after the last dose of study drug (refer to Appendix 6).
14. Concomitant use of any medications or substances that are strong inducers of CYP3A4 are prohibited within 21 days prior to randomization and during study treatment (refer to Appendix 6).
15. Has received (within the past 30 days or 5 × drug half-life prior to randomization, which is longer) or is expected to receive COVID-19 monoclonal antibody or convalescent COVID-19 plasma during study treatment.
16. Systemic glucocorticoid therapy (prednisone ≥ 20 mg/day or equivalent doses of other steroids) for at least 14 consecutive days within 30 days prior to randomization.
17. Has received any SARS-CoV-2 vaccine within 3 months prior to randomization.
18. Participating in another interventional clinical study with an investigational compound or device, including those for COVID-19.
19. Previous administration with any investigational drug or vaccine within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) prior to randomization.
20. Known prior participation in this trial or other trial involving SIM0417.
21. Women who are breastfeeding or have a positive pregnancy test in the pre-dose examinations. The following female patients who have documentation of either a or b below do not need to undergo a pregnancy test in the pre-dose examinations:

    1. Postmenopausal women (defined as cessation of regular menstrual periods for 12 months or more, and confirmed by a follicle-stimulating hormone test if <60 years old)
    2. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation
22. Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments.

    For subjects who have conditional ECG at screening only:
23. Clinically relevant or significant electrocardiographic abnormalities (e.g., second-degree type II AV block, left bundle branch block, etc.), including electrocardiographic QT interval corrected for heart rate using Fridericia 's correction formula (QTcF = QT/(RR0.33)) > 450 ms (males) or > 470 ms (females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Time to sustained recovery of 11 COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 (absence or return to the status before the onset) for two consecutive days.(Participant-completed study diary (COVID-19 symptoms and signs, and global impression questions))

SECONDARY OUTCOMES:
Time to sustained recovery of 5 COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when 5 COVID-19 symptoms get scores of 0 (absence or return to the status before the onset) or 1 (mild) for two consecutive days.
Time to sustained alleviation of 7 COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when 7 COVID-19 symptoms get scores of 0 (absence or return to the status before the onset) or 1 (mild) for two consecutive days.
Time to sustained alleviation of 11 COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 (absence or return to the status before the onset) or 1 (mild) for two consecutive days.
Viral load | Baseline through Day 14
  Changes of viral load compared to the baseline.
SARS-CoV-2 RNA | Baseline through Day 14
  Proportion of participants with SARS-CoV-2 RNA below the threshold.
Severe COVID-19 disease | Baseline through Day 29
  Incidence of disease progression by COVID-19 severity.
Hospitalization or death | Baseline through Day 29
  Proportion of participants with hospitalization or death from any cause.
ICU stay | Baseline through Day 29
  Proportion of participants admitted into ICU.
Requiring supplemental oxygen | Baseline through Day 29
  Proportion of participants requiring supplemental oxygen (low-flow nasal cannula, simple face mask).
Requiring mechanical ventilation/ECMO | Baseline through Day 29
  Proportion of participants requiring mechanical ventilation/ECMO.
Death (all cause) | Baseline through Week 12
  Proportion of participants with death (all cause).
WHO clinical progression scale score | Baseline through Day 29
  Change from baseline in WHO clinical progression scale score.
Time to sustained recovery of each targeted COVID-19 symptom | Baseline through Day 29
  The time from the start of treatment to the time when each targeted COVID-19 symptom gets scores of 0 (absence or return to the status before the onset) for two consecutive days.
Proportion of sustained recovery of COVID-19 symptoms | Baseline through Day 29
  Proportion of patients whose symptoms has been sustainedly recovered.
Severity of COVID-19 symptoms | Baseline through Day 29
  Severity of each COVID-19 symptom.
Composite symptom score | Baseline through Day 29
  Change from baseline in composite symptom score.
Treatment-Related Adverse Events (TEAEs) | Baseline through Day 29
  Incidence of Treatment-Related Adverse Events (TEAEs).
Serious Adverse Events (SAEs) | Baseline through Week 12
  Incidence of Serious Adverse Events (SAEs) Assessed.
The plasma concentration of SIM0417 | Baseline through Day 5
  The trough concentrations of SIM0417.

OTHER OUTCOMES:
Time to cessation of SARS-CoV-2 viral shedding (Viral load assessment) | Baseline through Day 29
  The length of time from the start of treatment to first time when the virus RNA is below the defined threshold.
Hospital and ICU stay | Baseline through Week 12
  Number of days in hospital and ICU stay in participants with COVID-19 related hospitalization.
COVID-19 related medical visits | Baseline through Day 29
  Number of COVID-19 related medical visits other than hospitalization.
WHO clinical progression scale | Baseline through Day 29
  Proportion of participants at each clinical status as assessed by WHO clinical progression scale.
Resolution of fever | Baseline through Day 29
  Time to resolution of fever (Defined as the time between the initiation of the study treatment and the resolution of fever).
Global Impression Questions | Baseline through Day 29
  Time to self-reported return to usual (pre-COVID-19) health status (Global Impression Questions, section 8.1.1).
Health Economic Outcome | Baseline through week 12
  Change from baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) index score at applicable timepoint; The EQ-5D-5L index score comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
viral variants | Baseline through Day 29
  Explore the prevalence of viral variants.
drug-resistance mutation | Baseline through Day 29
  Explore the clinical drug-resistance mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Principal Investigator — China-Japan Friendship Hospital
Locations (35):
- China (35):
  - Hefei First People's Hospital, Hefei, Anhui
  - Beijing Ditan Hospital Captial Medical University, Beijing, Beijing Municipality
  - Chongqing Public Health Medical Center, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangzhou Eighth People's Hospital Guangzhou Medical University, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - GuiZhou Province People's Hospital, Guiyang, Guizhou
  - Haikou people's Hospital, Haikou, Hainan
  - Hainan Third People's Hospital, Sanya, Hainan
  - Mudanjiang Kangan Hospital, Mudanjiang, Heilongjiang
  - Wuhan Jinyintan Hospital, Wuhan, Hubei
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - ZhongDa Hospital SouthEast University, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Xuzhou Infectious Disease Hospital, Xuzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Sixth People's Hospital of ShenYang, Shenyang, Liaoning
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Public health clinical center of Chengdu, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin first center hospital, Tianjin, Tianjin Municipality
  - Affliated Hangzhou XiXi Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - HwaMei Hospital University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Yao B-F, Yang Y, Xu S-S, Tang B-H, Chen J, Guo Z-J, Hu H-L, Zhang W, Fu S-M, Zhang X-F, Hao G-X, Yang X-M, Song L-L, Ye P-P, Liu L, Zhu S-W, Zheng Y, Zhao W. Model-informed drug development in public health emergency of international concern: accelerating marketing authorization of simnotrelvir. Antimicrob Agents Chemother. 2025 Nov 5;69(11):e0061425. doi: 10.1128/aac.00614-25. Epub 2025 Sep 18. PMID 40965470
- [Derived] Cao B, Wang Y, Lu H, Huang C, Yang Y, Shang L, Chen Z, Jiang R, Liu Y, Lin L, Peng P, Wang F, Gong F, Hu H, Cheng C, Yao X, Ye X, Zhou H, Shen Y, Liu C, Wang C, Yi Z, Hu B, Xu J, Gu X, Shen J, Xu Y, Zhang L, Fan J, Tang R, Wang C. Oral Simnotrelvir for Adult Patients with Mild-to-Moderate Covid-19. N Engl J Med. 2024 Jan 18;390(3):230-241. doi: 10.1056/NEJMoa2301425. PMID 38231624